CLINICAL TRIAL: NCT05594472
Title: Ozonated Olive Oil in Treatment of Pemphigus Vulgaris and Bullous Pemphigoid Compared to Conventional Topical Treatment
Brief Title: Ozonated Olive Oil in Treatment of Pemphigus Vulgaris and Bullous Pemphigoid
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rania Mogawer, Consultant and lecturer of dermatology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N-63-2021
Record Dates: First submitted 2022-10-21; First posted 2022-10-26 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Pemphigus Vulgaris; Bullous Pemphigoid
Keywords: Ozonated olive oil; Healing; Disinfection
MeSH Terms: conditions — Pemphigus; Pemphigoid, Bullous

STUDY DESIGN:
Intervention Model Description: A self controlled study on 2 contralateral comparative skin lesions
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ozonated olive oil (Experimental): ozonated oil will be applied to on one lesion followed by gauze for 5 consecutive days.
  Interventions: Drug: Ozonated olive oil
- Topical garamycin cream (Active Comparator): conventional topical treatment will be applied to a comparable lesion followed by gauze for 5 consecutive days.
  Interventions: Drug: Topical garamycin cream

INTERVENTIONS:
Drug: Ozonated olive oil — Topical treatment will be applied for 5 consecutive days on the erosions.
  Arms: Ozonated olive oil
Drug: Topical garamycin cream — Conventional topical treatment will be applied for 5 consecutive days on a comparable erosion
  Arms: Topical garamycin cream

SUMMARY:
This study assesses the disinfectant and healing promoting effect of ozonated olive oil in treatment of pemphigus vulgaris and bullous pemphigoid in comparison to conventional topical treatment with topical antibiotic.

DETAILED DESCRIPTION:
All participants will be subjected to the following:

* Written informed consent.
* Detailed history and clinical examination and photographic documentation
* Patients with pemphigus vulgaris (epidermal skin blisters) as well as those with bullous pemphigoid (subepidermal skin blisters) will receive systemic treatment, namely; pulse steroid therapy and either mycophenolate mofetil or azathioprine

  +/- monthly IV cyclophosphamide.
* Two comparable contralateral lesions will be selected in every patient, which will be randomly assigned to either ozonated oil or conventional treatment.
* Patients will apply ozonated oil to on one lesion followed by gauze compared to conventional topical gentamycin and potassium permanganate followed by gauze on the contralateral lesion. Role of topical treatment is essentially to prevent / treat secondary bacterial infection of skin erosions as well as promote wound healing by maintaining moist clean environment.
* Surface area of both lesions will be calculated using digital planimetry, prior to starting treatment and by the end of treatment; namely end of the first cycle of intravenous pulse steroids on day 6 which defines end of intervention. Percent reduction on either side will be calculated.
* For assessing disinfectant effect, swabs will be taken from the 2 selected lesions at the same intervals for assessing for bacterial as well as fungal growth.
* Patients with positive cultures for bacterial growth will be given systemic antibiotics according to culture and sensitivity

ELIGIBILITY:
Inclusion Criteria:

Pemphigus vulgaris or Bullous pemphigoid with bilateral skin erosions.

Exclusion Criteria:

- Age < 18 years . Pregnant/ lactating females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Healing promoting effect of ozonated olive oil | 5 days per patient
  comparing percent change in surface area by digital planimetry in 2 selected comparable lesion

SECONDARY OUTCOMES:
Disinfectant effect of ozonated olive oil | 5 days per patient
  Comparing incidence of bacterial and fungal growth in the 2 arms

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed El-Shazly, MD, Study Chair — Faculty of pharmacy, Ain Shams University
Locations (1):
- Dermatology Department, Cairo University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Participants' data that underlie reported results will be shared upon request, after deidentification
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and up to 12 months after article publication.
Access Criteria: Controlled Access:
  Researchers who provide a methodologically sound proposal will be allowed to access data to achieve aims in the approved proposal.